CLINICAL TRIAL: NCT04550845
Title: Understanding of Genetics by Men at Risk for Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ewan Cobran, Ph.D., Senior Associate Consultant, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 22-011303; K01CA230193 (NIH); NCI-2023-05978 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Genetic Literacy; Heath Communication; Focus Group Discussions; Prognostic Genomics Technology
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prostate Cancer Genetic Literacy Application (PCGLA) Educational Video. (Experimental): Focus group discussions about the PCGLA educational video post-study. Focus group audiotapes will be transcribed verbatim, and then entered into the qualitative data software package, NVivo 14. A data dictionary will be created for each technical term to establish acceptable and unacceptable responses. Trained coders will evaluate comprehension of the technical terms independently and then resolve disagreement by consensus.
  Interventions: Behavioral: Focus group analyses
- Prostate Cancer Genetic Literacy Application (PCGLA) Educational Video plus Communication Coaching. (Experimental): Focus group discussions about the PCGLA educational plus nurse-navigated, tailored, prostate cancer education and communication coaching post-study.
  Focus group audiotapes will be transcribed verbatim, and then entered into the qualitative data software package, NVivo 14. A data dictionary will be created for each technical term to establish acceptable and unacceptable responses. Trained coders will evaluate comprehension of the technical terms independently and then resolve disagreement by consensus. post-study. Focus group audiotapes will be transcribed verbatim, and then entered into the qualitative data software package, NVivo 14. A data dictionary will be created for each technical term to establish acceptable and unacceptable responses. Trained coders will evaluate comprehension of the technical terms independently and then resolve disagreement by consensus.
  Interventions: Behavioral: Focus group analyses

INTERVENTIONS:
Behavioral: Focus group analyses — Focus group audiotapes will be transcribed verbatim, and then entered into the qualitative data software package, NVivo 14 for analysis.

SUMMARY:
With this greater certainty regarding prognosis, men with localized prostate cancer are now equipped with make better treatment planning decisions. This study is designed to investigate the understanding of prognostic genetic technology in African American and rural White men at risk for localized prostate cancer.

DETAILED DESCRIPTION:
Novel genomic technology, such as microarray analyses and next-generation sequencing, have improved the understanding of prostate cancer biology and prognosis. The National Comprehensive Cancer Network (NCCN), in 2016, recommended that patients and clinicians consider tissue-based genetic tests for localized prostate cancer. However, while much enthusiasm currently exits for the rapidly increasing field of genomic medicine, the use of multi-gene mRNA expression panels raises the potential for further divergence in prostate cancer treatment outcomes by race and low socioeconomic status. We know that health disparities persist in low income groups despite the existence of evidence-based guidelines and that adoption of state-of-the-art methods often lag behind in these groups.

The goals of this study are to explore how men at risk for localized prostate cancer comprehend prognostic genetic technology, and examine how an educational video about genetics impacts patient-caregiver communication of prognostic genetic technology. The study rationale is that without direct attention to genomic comprehension, the enthusiasm that exists in the rapidly increasing field of prostate cancer genomic medicine may not translate into health benefits for men with localized prostate cancer. The central hypotheses are men with lower levels of education will demonstrate a severe lack of genomic comprehension of tissue-based genetic tests for localized prostate cancer; and tailored prostate cancer education will significantly improve communication in a low literacy population.

The study approach is innovative because it applies a mixed-methods community-engagement research framework to explore how African American and rural White men at risk for localized prostate cancer, comprehend and interpret data generated from genetic technology. The proposed research is significant because of its potential to improve public health by improving the understanding of prognostic genetics in minority, low income, and rural populations, and engage and educate these diverse communities about genomics.

ELIGIBILITY:
Inclusion Criteria:

* African-American or White men
* Living in a rural or urban areas
* Age 40 to 95 years old
* Able and willing to provide informed consent
* English-speaking
* Willing to participate in the study.

This study will use the United States Department of Agriculture Office of Rural Development's definition of rural, which is as a city or town that has a population less than 50,000 inhabitants to define rural.

This study will use the United States Census Bureau's definition of urban, which is a city or town that has a population greater than 50,000 inhabitants to define urban.

Exclusion Criteria:

Women will be excluded from participating in this study. However, women will be recruited to serve on an advisory panel to review the video-based educational tool for the comprehension of genomic terminology for prognostic genetic testing in patients with localized prostate cancer.

Ages: 40 Years to 95 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 90 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-09-27 (Estimated); Study Completion 2027-09-27 (Estimated)

PRIMARY OUTCOMES:
Estimate Genetic Literacy | Baseline
  The Rapid Estimate of Adult Literacy in Genetic - Short Form: An 8-item measure to asses adult literacy in genetics will be used.
Estimate Genetic Literacy | Pre-intervention
  The Rapid Estimate of Adult Literacy in Genetic - Short Form: An 8-item measure to asses adult literacy in genetics will be used.
Estimate Genetic Literacy | Immediately after the intervention
  The Rapid Estimate of Adult Literacy in Genetic - Short Form: An 8-item measure to asses adult literacy in genetics will be used.
Prostate Cancer Genetic Understanding | Baseline
  The Prostate Cancer Genetic Literacy Application (PCGLA) Educational Video, which was developed for this research, will be used as the study educational intervention. Prostate Cancer Genetic understanding will be assess with an 18-item knowledge prostate cancer genetic survey. The items are True or False.
Focus Group Discussion | Baseline
  A semi-structured focus group discussion about the Prostate Cancer Genetic Literacy Application (PCGLA) educational video.
Focus Group Discussion | Immediately after the intervention
  A semi-structured focus group discussion about the Prostate Cancer Genetic Literacy Application (PCGLA) educational video.

SECONDARY OUTCOMES:
Prostate Cancer Knowledge Scale | Baseline
  The Prostate Cancer Knowledge Scales a 12-item self-report measure developed to assess men's knowledge of prostate cancer risk factors, symptoms, prevention, screening, and treatment. Response options were multiple choice or true/false with each question also including an I don't know response option. Scoring was based on the percentage of questions answered correctly and ranged from 0 to 100.
Prostate Cancer Knowledge Scale | Pre-intervention
  The Prostate Cancer Knowledge Scales a 12-item self-report measure developed to assess men's knowledge of prostate cancer risk factors, symptoms, prevention, screening, and treatment. Response options were multiple choice or true/false with each question also including an I don't know response option. Scoring was based on the percentage of questions answered correctly and ranged from 0 to 100.
Prostate Cancer Knowledge Scale | Immediately after the intervention
  The Prostate Cancer Knowledge Scales a 12-item self-report measure developed to assess men's knowledge of prostate cancer risk factors, symptoms, prevention, screening, and treatment. Response options were multiple choice or true/false with each question also including an I don't know response option. Scoring was based on the percentage of questions answered correctly and ranged from 0 to 100.
Demographic Characteristics | Baseline
  Patients will be asked ended-questions to assess (1) race, (2) age, (3) marital status, (4) employment status, (5) current and/or past prostate cancer diagnoses, (6) occupation, (7) level of education, and 8) income.

CONTACTS AND LOCATIONS:
Overall Officials: Ewan K Cobran, PhD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials